CLINICAL TRIAL: NCT07346274
Title: Intra-operative Hypotension and Post-operative Lactate Level After Pancreatic-duodenectomy. A Prospective Multicenter Observational Study (HYPOL Study)
Brief Title: Intra-operative Hypotension and Post-operative Lactate Level After Pancreatic-duodenectomy.
Acronym: HYPOL
Status: Enrolling by invitation | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, mtedeschi, Istituto Clinico Humanitas
Other Study IDs: HYPOL; HYPOL (Registry Identifier: HYPOL)
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Serum Lactate Post-pancreatic Duodenectomy
Keywords: serum lactate; blood pressure; hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days

GROUPS / COHORTS (1):
- patients undergoing pancreatic duodenectomy

SUMMARY:
Intraoperative hypotension is a frequent occurrence during pancreaticoduodenectomy (PD) and has been associated with impaired tissue perfusion and organ dysfunction. However, its specific relationship with early postoperative hyperlactatemia and clinical outcomes in PD patients remains poorly characterized.

Identifying a correlation between time-weighted average hypotension (TWA65) and postoperative lactate levels could provide valuable insights for optimizing intraoperative hemodynamic management and improving postoperative outcomes in high-risk abdominal surgery.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the association between intraoperative hypotension, defined as TWA65 > 0.2 mmHg, and postoperative lactate levels (>2 mmol/L at RR0 and RR1), as well as lactate clearance. Secondary objectives include assessing the relationship between hyperlactatemia (>4 mmol/L), impaired lactate clearance (Lacclear < 0), and the incidence of postoperative complications. The study also investigates how intraoperative factors such as fluid balance, body temperature, duration of surgery, cardiac index (CI), and cardiac power index (CPI) affect lactate levels and clearance. The primary endpoints are postoperative lactate levels and lactate clearance, while secondary endpoints include hyperlactatemia, lactate clearance deficit, and their association with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years
* Undergoing open pancreaticoduodenectomy (DCP)

Exclusion Criteria:

* Age under 18 or over 85 years
* Severe cardiac disease classified as NYHA class III-IV
* Cirrhotic liver disease
* Pregnancy
* Puerperium or breastfeeding
* ASA (American Society of Anesthesiologists) physical status score greater than 3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open pancreaticoduodenectomy (PD), aged 18-80
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
hypotensive events | 1 hour post operative
  The primary objective of the study is to evaluate the association between intraoperative hypotension, defined as TWA65 > 0.2 mmHg, and postoperative lactate levels (>2 mmol/L at RR0 and RR1), as well as lactate clearance.

SECONDARY OUTCOMES:
serum lactate | 7 days
  assessing the relationship between hyperlactatemia (>4 mmol/L), impaired lactate clearance (Lacclear < 0), and the incidence of postoperative complications.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Humanitas Research Hospital, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No